CLINICAL TRIAL: NCT02489929
Title: Evaluation of Cytidine Deaminase for Patient Suffering of a Myelodysplasic Syndrom or an Acute Myeloid Leukemia and Treated by Azacytidine
Brief Title: Evaluation of Cytidine Deaminase for Patient Suffering of a Myelodysplastic Syndrom or an AML Treated by Azacytidine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01797-40
Record Dates: First submitted 2015-05-28; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes | interventions — Blood Specimen Collection; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient suffering of MDS or Myeloid leukemia (Experimental): The patients suffering of MDS or Acute myeloid leukemia will be the object of 8 sampling of blood (on tube EDTA) distributed as this: the first day of the usual treatment (azacytidine) at T0, T30 MIN, T60 MIN, T90 MIN, T120 MIN, then a second series of taking in the 5th day of treatment at T0, T30 MIN, T90 MIN to determine cytidine deaminase (CDA) activities by following its plasmatic dosage
  Interventions: Other: blood samples; Drug: azacytidine

INTERVENTIONS:
Other: blood samples — This clinical study aims at correlating the values in CDA levels with the risk of drug-related toxicities and to the clinical response to azacytidine treatment for patient suffering of MDS or Myeloid leukemia
Drug: azacytidine

SUMMARY:
Myelodysplastic syndrome (MDS) is a group of medical conditions derived from progressive bone marrow failure that result in ineffective production of blood cells. Depending on the severity, MDS reduces the quality of life to the point of being life-threatening. There is a probability of death at all stages of the disease, due to complications and co-morbidities, with progression to acute myeloid leukemia (AML) being the worst evolution. Azacytidine is a nucleosidic analog with original epigenetic mechanism of action that is widely used for treating a variety of myelodysplasic syndromes. Although generally well tolerated, severe and sometimes life-threatening toxicities were unexpectedly observed in some patients. Genetic polymorphism affecting cytidine deaminase (CDA), the liver enzyme responsible for azacytidine detoxification step, could be responsible for poor clinical outcome due to on the one hand to severe toxicities in deficient patients, and on the other hand on treatment failure in ultrametabolizer patients.This clinical study aims at correlating the values in CDA levels with the risk of drug-related toxicities and to the clinical response to azacytidine treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients have to be capable of submitting themselves at the rate of the visits, in the plan of treatmen, in the balance assessments of laboratory and other procedures of the study.
* Patient treated by azacytidine

Exclusion Criteria:

* Patients having an infection unchecked who could compromise the participation in the study
* Patients having other grave and/or unchecked concomitant diseases which could compromise the participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of survival without progress of the disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Regis COSTELLO, MD, Principal Investigator — AP-HM
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France